CLINICAL TRIAL: NCT04105049
Title: Multivariate Predictive-discriminatory Model of Academic Performance in Medical Students. A Mixed Longitudinal Study.
Status: Completed | Type: Observational
Sponsor: Raúl Sampieri Cabrera (Other)
Responsible Party: Sponsor-Investigator, Raúl Sampieri Cabrera, Master of Science, Associate Professor B TC, Universidad Nacional Autonoma de Mexico
Organization: Universidad Nacional Autonoma de Mexico (Other)
Other Study IDs: IN309920
Record Dates: First submitted 2019-08-26; First posted 2019-09-26 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Students at Risk of Obtaining Low Academic Performance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation of psychological aspects — Motivational, socioeconomic, family, stress, and other aspects are tested.

SUMMARY:
Reported studies on individual differences related to academic performance based on personality aspects describe self-efficiency, motivation and self-control as the main indicators of academic performance. Students who are motivated tend to have a better academic performance (AP) than peers with less motivation. On the other hand, differences in the environment related to academic performance have been linked to social aspects, among which are: family environment, family socioeconomic status and academic socialization. A constant factor in aspects of the environment that seems to permeate and impose itself on others is the socioeconomic one. About the personal factors of medical students, it has been found that university students who report stress caused by socioeconomic factors are more likely to have some psychological morbidity. There are certain ways to deal with stress that are related to better performance. Due to the complexity of the study of AP, it is necessary to develop holistic models that allow a better approach to reality. The educational research work related to academic disillusionment has been aimed at determining the factors involved in it. However, the methodological approach that has been used to document these works focuses on reductionism, where each variable that is studied and correlated independently with the AP. Although, this approach has provided valuable information, it is necessary to postulate holistic models that allow a better approach to reality. Although, there are published works on the correlation of the factors that can influence the academic performance of medical students of the Faculty of Medicine of the UNAM, no multivariate predictive models have been developed that include the main psychosocial factors and the resilience of students and how they impact academic performance; and also, study their behavior throughout a school year of the career, using stochastic models that allow characterizing a succession of random variables that evolve as a function of time. Therefore, the present work has as main purpose to establish a predictive model that allows predictions of expected academic performance and timely detection of students in situations of academic risk; and in turn tutorials, educational guidance, psychological support and / or specialized advice.

DETAILED DESCRIPTION:
The medical career demands of its students a great dedication and dedication, which for some can become a problem that leads to an alteration of the state of physical and mental health. Those who have dedicated themselves to studying academic performance and its impact on mental health point out that the stress, anxiety and depression experienced by students throughout the school year are factors that cause poor academic performance (AP). The AP is defined as the degree to which a student has achieved educational goals satisfactorily. It is usually measured through tests or continuous evaluations. Individual differences related to academic performance have been linked to cognitive and personality aspects (non-cognitive skills). In cognitive aspects, it has been reported that students with a higher IQ and those who have greater awareness of effort and achievement tend to have high performance in academic settings. In addition, it has also been suggested that mental curiosity (measured by intellectual commitment) has an important influence on academic achievement. In relation to personality aspects, understood as a set of "attitudes, behaviors and strategies" that promote academic and professional success. It has been reported that academic self-efficiency, self-control, motivation, expectation and goal-setting theories, emotional intelligence and determination are non-cognitive skills that provide a better explanation of AP. Reported studies on individual differences related to academic performance based on personality aspects describe self-efficiency, motivation and self-control as the main indicators of academic performance. Self-efficacy is understood as an individual's belief that he can do something. Stajković and collaborators demonstrated that self-efficacy is one of the best predictors of academic success. In addition, they reported that emotional awareness and stability were predictors of self-efficacy; Students who are motivated tend to have better academic performance than peers with less motivation; and self-control, in the academic environment, is related to self-discipline, self-regulation, delay of self-gratification and impulse control. That is, self-control is the ability to prioritize long-term objectives over the temptation of short-term impulses. On the other hand, differences in the environment related to academic performance have been linked to social aspects, among which the following stand out: family environment, family socioeconomic status and academic socialization. In the family environment it has been described that the quality of the relationship between parents and students influences the development of academic self-efficacy, which in turn will contribute to their AP; With regard to family socioeconomic status it has been reported that students of parents with lower economic incomes lack an academic environment at home, which influences their academic success. In particular, books at home have been associated as one of the most influential factors in student performance, in addition, highly educated parents (who have improved their family income) tend to have learning environments more stimulants; Academic socialization is understood as the interaction that the student establishes with classmates and academic-administrative staff, studies have linked it to the development of extracurricular activities, which have resulted in positive relationships between students and high performance. academic which includes the increase of the rates of attendance to classes, greater school commitment, as well as a decrease in the rates of abandonment and depression or student frustration. Among the most studied extracurricular activities is physical exercise that has been shown to improve academic performance in university students, in addition to increasing neuronal activity in the brain, especially the increase in executive brain functions, such as attention span and working memory. A constant factor in aspects of the environment and that seems to permeate and impose itself on others is the socioeconomic one, where it has been described that academic socialization can be influenced by family socioeconomic status. The socioeconomic level also impacts education institutions, in the report Coleman concluded that students who attend a school in which the average socioeconomic level is high enjoy better educational results compared to one where, the students have a low socioeconomic level. From the beginning, parents with a higher socioeconomic status can provide students with financial support and household resources for individual learning.

Regarding the personal factors of medical students, it has been found that university students who report stress caused by socioeconomic factors are more likely to have some psychological morbidity. One possible explanation is that the entrance to the university and the academic difficulties represent a set of stressful situations that can generate a temporary emotional lack of control in the students. A diagnostic test is applied at the Faculty of Medicine of the UNAM; in which several areas of conceptual auscultation are evaluated, it has been shown that the academic background of the baccalaureate play a very important role in the level of accreditation that is reached in the different subjects of the medical career. On the other hand, there are certain ways to deal with stress that are related to better performance. Due to the complexity of the study of AP, it is necessary to develop holistic models that allow a better approach to reality. Therefore, this work has as main purpose to establish predictive models that allow predictions of expected academic performance and timely detection of students in situations of academic risk; and in turn tutorials, educational guidance, psychological support and / or specialized counseling. In addition, due to the complex nature of the phenomenon, a qualitative study will be carried out using phenomenological methodology, which will explore specific social aspects that could be imperceptible in quantitative tests.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female students of the Department of physiology of the Faculty of Medicine of the National Autonomous University of Mexico
2. Voluntarily accept your participation in the study by signing the informed consent.

Exclusion Criteria:

1. Students who have difficulty or refuse to fill the scales
2. Students who withdraw their informed consent at any time during the study

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be carried out in the Department of Physiology of the Faculty of Medicine of the National Autonomous University of Mexico during the 2019-2020 school year.
  Selection criteria.
  In January 2019, physiology students will be informed and invited to participate personally after authorization of the head teacher of each group, explaining the voluntary nature of the study, the nature of the study and the student's participation in it.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
academic performance | 3 years
  Numerical qualification of the subjects of the second year of medicine of the School of Medicine of the UNAMnumerical qualification of the subjects of the second year of medicine of the Faculty of Medicine of the UNAM

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Inclán-Rubio, PhD, Principal Investigator — Facultad de Medicina, UNAM
Locations (1):
- Departamento de Fisiología, Facultad de Medicina, UNAM, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided